CLINICAL TRIAL: NCT01693926
Title: Effect of Physical Activity an Stress in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Jardena Puder, Medin adjoint, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 286/12
Record Dates: First submitted 2012-08-29; First posted 2012-09-26 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Children; Physical Activity; Stress; Snacking
Keywords: Obesity; Children; Physical activity; Stress; Snacking
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute physical activity intervention (Experimental): 25 min of moderate physical activity
  Interventions: Behavioral: Acute physical activity intervention
- Placebo (Placebo Comparator): 25 min of reading (instead of physical activity)
  Interventions: Behavioral: placebo

INTERVENTIONS:
Behavioral: Acute physical activity intervention — 25 min of physical activity. The placebo arm will have 25 min of reading.
  Arms: Acute physical activity intervention
Behavioral: placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the impact of physical activity in obese and nonobese prepubertal children on:

1. biological stress responses during a psychosocial stress test
2. snacking and feeling of hunger in response to the same psychosocial stress test
3. the moderating factor of attachment on the biological stress responses and on snacking

Children will be investigated on one study day during 3.5 hours.

DETAILED DESCRIPTION:
Hypotheses In this study, 3 primary hypotheses will be tested.

1. Moderate physical activity during 25 min in children decreases the cortisol levels in response to the Trier Social Stress Test TSST-C (for children).
2. Moderate physical activity during 25 min in children decreases the snacking (calorie consumption when corrected for expenditure and switch in quality of food intake) in response to the Trier Social Stress Test TSST-C (for children).
3. A secure attachment will be a moderating factor for the general increase in cortisol and the snacking in response to the psychosocial stress test (Trier Social Stress Test TSST-C).

Secondary objectives:

1. To test if the impact of physical activity on stress responses and snacking differs between obese and non-obese children
2. To test the impact of physical activity on the cardiovascular stress reactivity (blood pressure, heart rate) and the perceived stress (scale) in response to the Trier Social Stress Test TSST-C?
3. To test if the stress reactivity and its modulation by physical activity is different in anxious and in impulsives/labile children
4. To test if serious life events and parental worries and parental educational style influence the stress reactivity

ELIGIBILITY:
Inclusion Criteria:

* 7-10 year old children

Exclusion Criteria:

* Severe illness
* Medications interfering with study

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in salivary Cortisol and maximal levels of salivary cortisol in response to the TSST stress test over 2 hours | 9 months
Snacking (Caloric intake, corrected for energy expenditure) | 9 months
  Measure of caloric intake and measure of choice of high-caloric vs low-caloric food snacking after the TSST stress test
Moderator effect of attachment (4 different attachment categories), i.e. children with a secure attachment will have lower rises in cortisol compared with children in the other 3 attachment categories | 9 months
  Cortisol levels after the TSST stress test will be lower in children with secure attachment compared to detached, disorganized or preoccupied children (i.e. the 3 other attachment categories).

SECONDARY OUTCOMES:
Moderator effect of obesity (WHO criteria) | 9 months
Cardiovascular reactivity (changes and maximal levels of blood pressure, heart rate) | 9 months
Perceived stress (stress scale from 1-7) | 9 months
Moderator role of serious life events and parental worries | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Lausanne, SUPEA, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Horsch A, Wobmann M, Kriemler S, Munsch S, Borloz S, Balz A, Marques-Vidal P, Borghini A, Puder JJ. Impact of physical activity on energy balance, food intake and choice in normal weight and obese children in the setting of acute social stress: a randomized controlled trial. BMC Pediatr. 2015 Feb 19;15:12. doi: 10.1186/s12887-015-0326-7. PMID 25879821